CLINICAL TRIAL: NCT05438004
Title: NICE BIRTH - Ambulatory Childbirth Pathway Pilot Feasibility Study
Brief Title: Ambulatory Childbirth Pathway Pilot Feasibility Study
Acronym: NICE BIRTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-PP-10
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related
Keywords: Ambulatory; Childbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulatory nice birth (Experimental): Discharge from the maternity ward from the 2nd hour and before the 24th hour following an uncomplicated delivery
  Interventions: Other: Ambulatory nice birth

INTERVENTIONS:
Other: Ambulatory nice birth — discharge from the maternity ward from the 2nd hour and before the 24th hour following an uncomplicated delivery

SUMMARY:
In 2016, according to the national perinatal survey, the average length of stay in maternity hospitals in France after a vaginal delivery was 4.0 days, confirming the decrease in this length of stay compared with previous surveys, but placing France among the Western countries with the longest stay.

Several countries that have further reduced the average length of stay offer low-risk populations a return home in the first few hours after delivery.

As early as 2014, the Haute Autorité de Santé reminded us that "once low risk is defined, the length of stay in the maternity hospital is not discriminating for the safety of the mother and the newborn. The optimal length of stay would rather depend on the organization of the discharge from the maternity hospital, the medical follow-up and the subsequent support".

The studies against a very early discharge are the result of experiments that do not define low risk, and/or do not propose home support.

This pilot study aims to provide a framework for a care pathway allowing discharge from the maternity hospital from the 2nd hour and before the 24th hour following an uncomplicated delivery. Its main objective is to show that such a care pathway allows to respect the French postpartum recommendations, while answering a legitimate expectation of personalization of the care offered to women wishing to be monitored at home earlier after the delivery. It also studies the complications, tolerance, satisfaction and cost of such care.

This is a non-randomized cohort study. It studies 100 voluntary mother-newborn couples, after a delivery at the Nice University Hospital, meeting objective criteria of low risk. A daily follow-up is ensured by a liberal midwife during the first 3 days. The link between the patient, the private midwife and the maternity hospital is maintained permanently thanks to a free dedicated mobile application. This application, equipped with an alert system, is an additional guarantee of compliance with the recommendations for screening and mandatory procedures. It allows for a safer transfer of hospital care to ambulatory care, while providing personalized care tailored to the patient's expectations.

This pilot study would be the beginning of a larger study demonstrating the non-inferiority of such a care pathway compared to the most common management requiring a stay of several days in a maternity hospital.

ELIGIBILITY:
Inclusion Criteria:

* Maternal:
* Voluntary
* Legal age
* Vaginal delivery
* General Health Insurance Plan
* Accompanying person present at discharge and every day during the first 2 days
* Pain VAS < 5 with or without simple analgesics
* Mother-child interaction judged satisfactory by the team
* Signature of consent
* Pediatric :
* Singleton
* > 38 weeks of amenorrhea
* Eutrophic
* Apgar > 7 at 5 minutes of life
* Respiratory rate < 60/min; 90bpm < Heart rate < 170bpm; SaO2 >95
* Axillary temperature between 36 and 37°C
* Feeding established
* Vitamin K1 given
* Neonatal screenings organized

Exclusion Criteria:

* Maternal:
* Social isolation, psychiatric disorder with impact on infant care, moderate to severe (according to DSM5) substance use disorder
* Poorly balanced chronic condition requiring hospitalization
* Postpartum complications requiring hospitalization
* Postpartum hemorrhage > 500mL
* Body temperature > 38.0°C without paracetamol
* Thromboembolic signs: pain, edema, positive Homans sign
* Protected persons defined in the following articles of the public health code:

L. 1121-6: persons deprived of liberty by a judicial or administrative decision, persons hospitalized without consent and persons admitted to a health or social institution for purposes other than research; L. 1121-8: adults subject to a legal protection measure or unable to express their consent; L. 1122-1-2: persons in emergency situations unable to give prior consent.

* Pediatric :
* Jaundice
* Risk factor for neonatal infection (maternal streptococcal B colonization during the current pregnancy, history of neonatal streptococcal B infection in a previous pregnancy, duration of rupture of membranes > 12 hours, maternal temperature > 38.0°C intrapartum or during the 2 hours following delivery).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Emergency visits | one month
  Percentage of emergency visits for neonatal or maternal reasons within one month of delivery

SECONDARY OUTCOMES:
post partum recommendations | one month
  Number of deviations from postpartum recommendations
Breastfeading rate | one month
  Difference between the breastfeeding desire rate on the day of delivery and the breastfeeding rate at 1 month postpartum
Maternal pain | Day 2
  Maternal pain on the 2nd day of delivery measured with the VAS scale, ranging from 1 (no pain) to 10 (maximum imaginable pain)
Satisfaction score | One month
  Overall satisfaction score for care at 1 month postpartum ranging from 1 (not satisfied) to 10 (very satisfied)
Cost of outpatient care | one month
  Average cost (in euros) of outpatient care: cost of shortened hospitalization + cost of consultations with the private midwife + cost of managing alerts from the remote application

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexis GAUCI, MD-PHD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Archet, Nice, France